CLINICAL TRIAL: NCT05423067
Title: Interventional Gynecologic Surgery
Brief Title: Permanent Occlusion of Uteine Arteies in Management of Abnormal Uterine Bleeding
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura Integrated Fertility Center (Other)
Responsible Party: Principal Investigator, Emad Mohamad Sedeek, professor, Mansoura Integrated Fertility Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adelhelal
Record Dates: First submitted 2015-12-09; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Other Abnormal Uterine and Vaginal Bleeding
Keywords: permenant occlusion; uterine bleeding; uterine arteries
MeSH Terms: conditions — Uterine Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BUAO (Other): The study done in two phases:
  1. Phase one from October 2011to May 2012 pilot study including twenty nine (29) premenopausal patients followed up for six months
  2. Phase two from October 2012 till May 2014. Including Eighty nine (89) premenopausal patients
  Interventions: Procedure: bilateral permanent occlusion of uterine arteries

INTERVENTIONS:
Procedure: bilateral permanent occlusion of uterine arteries — bilateral permanent Occlusion of uterine arteries through abdominal route

SUMMARY:
Prospective observational interventional study , The study done in two phases:

1. Phase one from October 2011to May 2012 pilot study including twenty nine (29) premenopausal patients followed up for six months
2. Phase two from October 2012 till May 2014. Including Eighty nine (89) premenopausal patients all of them needing to preserve their uteri.

DETAILED DESCRIPTION:
Abstract Objectives: To assess the effectiveness of permanent bilateral occlusion of uterine arteries in treatment of abnormal uterine bleeding.

Design: prospective observational study Setting: Done in Mansoura university hospital, department of Obstetrics and gynecology.

Patients and Methods: The study done in two phases:

1. Phase one from October 2011to May 2012 pilot study including twenty nine (29) premenopausal patients followed up for six months
2. Phase two from October 2012 till May 2014. Including Eighty nine (89) premenopausal patients all of them needing to preserve their uteri.

Results: Results are hopeful and courageous in phase one as regards patients satisfaction, Quality of life and improvements of bleeding. Results of phase two will be implemented, analyzed and presented in tables. All data will be statistically analyzed and the results will be presented after completion of eighteen (18) months follow up to rule out any bias and/ or errors in the results.

Conclusion: permanent bilateral uterine arteries occlusion may be a good alternative to radical surgery in abnormal uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal with abnormal uterine bleeding and completed their families having normal endometrium (biopsy in preceding 6 months ) and may have uterine intramural myomas not exceeding 150 ml in volume and away from uterine cavity by at least 1cm and /or adenomyosis

Exclusion Criteria:

* patients wishing future fertility
* endometrial sampling not done or more than 6 months or myoma encroaching or distorting cavity or larger than 150 ml in volume

Ages: 34 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
uterine bleeding | October 2011 till January 2016

SECONDARY OUTCOMES:
patient satisfaction | october 2011 - may 2015
quality of life | october 2011 - may 2015

CONTACTS AND LOCATIONS:
Overall Officials: Adel S Helal, MD, Principal Investigator — Mansoura Integrated Fertility Center
Locations (1):
- Mansoura Integrated fertility center, Al Mansurah, Dekahlia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided